CLINICAL TRIAL: NCT06997887
Title: Promotion of Vaginal Health With CH2 Vaginal Gel After Pelvic Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Jenny Ling-Yu Chen, MD PhD, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202503152RIPE
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Malignancy
Keywords: pelvic radiotherapy; CH2 vagina gel; vagina rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will undergo a 12-week intervention with either CH2 vaginal gel or vaginal rehabilitation exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CH2 vaginal gel (Experimental): Female patients who have completed pelvic radiotherapy, participants will undergo a 12-week intervention with CH2 vaginal gel.
  Interventions: Other: CH2 vaginal gel
- vaginal rehabilitation exercises (Active Comparator): Female patients who have completed pelvic radiotherapy, participants will undergo a 12-week intervention with vaginal rehabilitation exercises.
  Interventions: Other: vaginal rehabilitation exercises

INTERVENTIONS:
Other: CH2 vaginal gel — 12-week intervention with CH2 vaginal gel
  Arms: CH2 vaginal gel
Other: vaginal rehabilitation exercises — 12-week intervention with vaginal rehabilitation exercises
  Arms: vaginal rehabilitation exercises

SUMMARY:
This is a prospective clinical trial planning to enroll female patients who have completed pelvic radiotherapy. Participants will undergo a 12-week intervention with either CH2 vaginal gel or vaginal rehabilitation exercises. The primary endpoint is the change in the Female Sexual Function Index scores.

DETAILED DESCRIPTION:
This is a prospective clinical trial planning to enroll female patients who have completed pelvic radiotherapy. Participants will undergo a 12-week intervention with either CH2 vaginal gel or vaginal rehabilitation exercises. The primary endpoint is the change in the Female Sexual Function Index (FSFI) scores. Follow-up assessments will be conducted to determine whether CH2 vaginal gel or vaginal rehabilitation can improve post-radiotherapy vaginal health and enhance the long-term quality of life for women with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 20 and 70 years.
2. Completion of pelvic radiotherapy for gynecologic cancer, which may include external beam radiotherapy (EBRT), brachytherapy (BT), or a combination of both.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.

Exclusion Criteria:

1. Individuals under the age of 18.
2. Presence of distant metastases or a history of malignancy currently under treatment within the past five years (excluding non-melanoma skin cancer).
3. Presence of severe comorbidities, such as uncontrolled diabetes, cardiovascular disease, or autoimmune disorders that may interfere with treatment or study participation.
4. Diagnosed psychiatric disorders or significant social factors that may prevent adherence to study requirements or completion of follow-up evaluations.
5. Inability to self-administer vaginal gel or vaginal rehabilitation exercises.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2028-05-09 (Estimated); Study Completion 2030-05-09 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) score | From enrollment to the end of intervention at at 3, 6, and 12 months
  Female Sexual Function Index (FSFI) score. The score ranges from a minimum of 2 to a maximum of 36. Higher scores indicate better sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ling-Yu Chen Professor, Attending Physician, MD PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Patient privacy consideration.